CLINICAL TRIAL: NCT05752474
Title: Multi-Component Prehabilitation Program for High-Risk Older Adults Undergoing Major Elective Surgery: A Pilot and Feasibility Study
Brief Title: Multi-Component Prehabilitation for Major Elective Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Dae Hyun Kim, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000090
Record Dates: First submitted 2023-02-22; First posted 2023-03-02 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Frailty; Functional Recovery; Prehabilitation
Keywords: Prehabilitation; Surgery; Feasibility Studies
MeSH Terms: conditions — Frailty | interventions — Exercise; Nutritional Status; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation (Experimental): This group will receive a multicomponent prehabilitation intervention (exercise, nutritional intervention, meditation, and cognitive behavioral intervention) for 3-4 weeks prior to surgery.
  Interventions: Behavioral: Exercise; Behavioral: Nutrition; Behavioral: Meditation; Behavioral: Cognitive Behavioral Intervention

INTERVENTIONS:
Behavioral: Exercise — Physical therapy targeting flexibility, strength, and endurance will be delivered at the participant's home, center-based, or virtually via a twice-weekly (on average) schedule to provide a total of about 6-8 sessions during the 3-4 week study period. Participants will be asked to participate in self-directed exercise for at least 30 minutes per day for 4 or more days per week.
Behavioral: Nutrition — One-hour virtual group nutrition education classes will be held once per week by a dietitian, focusing on optimal protein intake (1.2 grams per kg of body weight) for lean body mass preservation (from food sources and oral nutritional supplements) and muscle gain. Participants will also receive oral nutritional supplements (20-30 grams of protein/day provided by our study team).
Behavioral: Meditation — One-hour virtual group meditation sessions will be held once per week by an experienced meditation teacher. Classes will focus on breathing techniques, yoga, and mindful meditation practices. Participants will be asked to participate in self-directed meditation for at least 12 minutes daily.
Behavioral: Cognitive Behavioral Intervention — A 30-min telephone-based session with individual patients will take place to deliver cognitive behavioral strategies once per week by a professionally trained clinician. These strategies include education about frailty and surgery, increasing positive beliefs of the benefits of exercise and nutrition, discussing barriers, setting individualized goals for surgery and recovery, developing a detailed exercise and nutrition plan (including logistics), self-monitoring of progress using weekly exercise, diet, and meditation logs, and enhancing self-efficacy through the celebration of small wins.

SUMMARY:
The purpose of this pilot study is to assess the feasibility of delivering a multicomponent prehabilitation and measuring patient-centered outcomes in older adults undergoing major surgery.

DETAILED DESCRIPTION:
We will assess the feasibility of delivering a multicomponent prehabilitation, which consists of exercise (supervised by physical therapist), nutritional intervention (nutritional supplement and group education), meditation (group class), and cognitive behavioral intervention over 3-4 weeks before major elective abdominal, gynecological oncologic, urologic surgery, and cardiovascular procedures. We will also measure patient-centered outcomes (Patient-Reported Outcomes Measurement Information System) at 30 and 90 days after surgery. The target enrollment is 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled to have a gastrointestinal, gynecological oncologic, urologic, and cardiovascular procedure
* Age 70 years+
* Age 65 years+ AND high risk per surgeon's clinical judgment
* Patient provides an informed e-consent or remote consent

Exclusion Criteria:

* Surgery is scheduled less than 21 days
* Patient is considered an inappropriate candidate per the surgeon's assessment
* Non-English speaking
* Major cognitive impairment
* Patients with chronic kidney disease stage 3 or higher will be excluded from receiving protein supplement of the prehabilitation program

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hyun Kim, MD, ScD, Principal Investigator — Beth Israel Deaconess Medical Center, 330 Brookline Ave, Boston, MA 02215
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Because this is a feasibility study of a multicomponent prehabilitation intervention, we do not plan to share individual participant data to other researchers.

REFERENCES:
- [Derived] Wang KY, Xu K, Liu Y, Alshanniek S, Newmeyer N, Mesnik L, Prudhivi V, Chase T, Rangasamy V, Sison SM, Shi SM, Travison TG, Subramaniam B, Kim DH. Multi-Component Prehabilitation Program for Older Adults Undergoing Major Elective Surgery: A Pilot and Feasibility Study. J Am Geriatr Soc. 2025 Nov;73(11):3387-3395. doi: 10.1111/jgs.70095. Epub 2025 Sep 7. PMID 40916355

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 patients were enrolled in the single-arm trial.
Groups:
- Prehabilitation: An Individualized, Multi-component Program: This single-arm trial was conducted at Beth Israel Deaconess Medical Center (enrollment site) and Hebrew Rehabilitation Center (intervention site) in Boston, Massachusetts, from March 2023 to January 2025. Patients 65 years or older scheduled for major abdominal, gynecological oncologic, urologic, and cardiovascular procedures were eligible. The program included the following components:
  1. Physical therapy: Participants received two one-hour individual sessions per week, delivered by a physical therapist at the Hebrew Rehabilitation Center.
  2. Nutrition: Participants received a one-hour individual nutritional counseling virtually by a registered dietitian. They were supplied with a protein bar or drink containing 20 grams of protein and instructed to consume daily, preferably within 30 minutes of exercise, to maximize muscle protein synthesis.
  3. Meditation: A meditation instructor at the Beth Israel Deaconess Medical Center Sadhguru Center for a Conscious Planet led a weekly one-hour virtual group meditation session. These sessions focused on breathing techniques and mindfulness practices to alleviate psychological stress, manage anxiety, and promote mental well-being.
Period: Overall Study
Arm/Group | Prehabilitation: An Individualized, Multi-component Program
Started | 30
Initiated Intervention (28 patients initiated the intervention.) | 28
Underwent Surgery (23 patients underwent surgery.) | 23
Completed | 21 (21 patients completed 90-day follow-up survey.)
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Prehabilitation: An Individualized, Multi-component Program
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Prehabilitation Program
Description: Measurement: Percentage of patients to whom we can deliver an adequate dose (≥50% of the planned sessions) of the 3 core interventions: physical therapy (≥4/8 sessions), nutrition (≥2/3-4 sessions), and meditation (≥2/3-4 sessions).
  Range: 0-100% (higher values indicate higher feasibility).
Time Frame: Post-intervention (up to 4 weeks)
Population: This was calculated in 28 patients who initiated the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Prehabilitation
Number analyzed (Participants) | 28
Participants | 19

2. Post Hoc Outcome: Change in Gait Speed
Description: Measurement: gait speed (meters/second) over 5-meter fast walk, post-intervention minus pre-intervention baseline Range: 0 to 2 meter/second Interpretation: Higher values indicate faster gait.
Time Frame: Between pre-intervention baseline and post-intervention (up to 4 weeks)
Population: This was calculated in 25 patients who initiated the intervention and had the post-intervention measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: meter/second
Arm/Group | Prehabilitation
Number analyzed (Participants) | 25
meter/second | 0.2 [0.0 to 0.4]

3. Secondary Outcome: Change in 5-chair Stand Test Time
Description: Measurement: Time to complete 5 chair stands (seconds), post-prehabilitation (up to 4 weeks) minus pre-prehabilitation baseline Range: 0 to 60 seconds Interpretation: Higher values indicate worse lower extremity strength.
Time Frame: Between pre-intervention baseline and post-intervention (up to 4 weeks)
Population: This was calculated in 25 patients who initiated the intervention and had the post-intervention measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Prehabilitation
Number analyzed (Participants) | 25
Seconds | -3.4 [-6.9 to 0.0]

4. Secondary Outcome: Change in Dominant Handgrip Strength
Description: Measurement: Average of 3 measurements of dominant handgrip strength (kilograms) measured using a Jamar dynamometer, post-prehabilitation (up to 4 weeks) minus pre-prehabilitation baseline Range: 0 to 60 kilograms Interpretation: Higher values indicate greater muscle strength
Time Frame: Between pre-intervention baseline and post-intervention (up to 4 weeks)
Population: This was calculated in 25 patients who initiated the intervention and had the post-intervention measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Prehabilitation
Number analyzed (Participants) | 25
Kilograms | 1.6 [-2.1 to 5.3]

5. Secondary Outcome: Adherence to Exercise
Description: Measurement: percentage of physical therapy sessions attended Range: 0-100% (higher values indicate better adherence)
Time Frame: Post-intervention (up to 4 weeks)
Population: This was calculated in 28 patients who initiated the intervention.
Measure: Count of Units; unit: Number of Sessions
Units Other Than Participants: Number of Sessions
Arm/Group | Prehabilitation
Number analyzed (Participants) | 28
Number analyzed (Number of Sessions) | 208
Number of Sessions | 190

6. Secondary Outcome: Adherence to Nutrition
Description: Measurement: percentage of nutrition sessions attended Range: 0-100% (higher values indicate better adherence)
Time Frame: Post-intervention (up to 4 weeks)
Population: This was calculated in 28 patients who initiated the intervention.
Measure: Count of Units; unit: Number of Sessions
Units Other Than Participants: Number of Sessions
Arm/Group | Prehabilitation
Number analyzed (Participants) | 28
Number analyzed (Number of Sessions) | 104
Number of Sessions | 80

7. Secondary Outcome: Adherence to Meditation
Description: Measurement: percentage of meditation sessions attended Range: 0-100% (higher values indicate better adherence)
Time Frame: Post-intervention (up to 4 weeks)
Population: This was calculated in 28 patients who initiated the intervention.
Measure: Count of Units; unit: Number of Sessions
Units Other Than Participants: Number of Sessions
Arm/Group | Prehabilitation
Number analyzed (Participants) | 28
Number analyzed (Number of Sessions) | 104
Number of Sessions | 71

8. Other Pre Specified Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS)-Computer Adaptive Test (CAT) Physical Function T Score
Description: Measurement: Self-reported measure of physical function, 90 days after surgery minus pre-intervention baseline Range: Standardized score with a mean of 50 and a standard deviation of 10 Interpretation: Higher scores indicate better physical function
Time Frame: Between pre-intervention baseline and 90 days after surgery
Population: This was calculated in 22 patients who initiated the intervention and had the 90-day measurement after surgery.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 22
score on a scale | 4.4 [3.0 to 5.9]

9. Other Pre Specified Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS)-Computer Adaptive Test (CAT) Anxiety T Score
Description: Measurement: Self-reported measure of anxiety, 90 days after surgery minus pre-intervention baseline Range: Standardized score with a mean of 50 and a standard deviation of 10 Interpretation: Higher scores indicate greater anxiety
Time Frame: Between pre-intervention baseline and 90 days after surgery
Population: This was calculated in 22 patients who initiated the intervention and had the 90-day measurement after surgery.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 22
score on a scale | -6.4 [-7.8 to -4.9]

10. Other Pre Specified Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS)-Computer Adaptive Test (CAT) Depression T Score
Description: Measurement: Self-reported measure of depression, 90 days after surgery minus pre-intervention baseline Range: Standardized score with a mean of 50 and a standard deviation of 10 Interpretation: Higher scores indicate more depressive mood
Time Frame: Between pre-intervention baseline and 90 days after surgery
Population: This was calculated in 22 patients who initiated the intervention and had the 90-day measurement after surgery.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 22
score on a scale | -2.6 [-3.7 to -1.5]

11. Other Pre Specified Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS)-Computer Adaptive Test (CAT) Fatigue T Score
Description: Measurement: Self-reported measure of fatigue, 90 days after surgery minus pre-intervention baseline Range: Standardized score with a mean of 50 and a standard deviation of 10 Interpretation: Higher scores indicate worse fatigue
Time Frame: Between pre-intervention baseline and 90 days after surgery
Population: This was calculated in 22 patients who initiated the intervention and had the 90-day measurement after surgery.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 22
score on a scale | -4.8 [-6.3 to -3.3]

12. Other Pre Specified Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS)-Computer Adaptive Test (CAT) Sleep Disturbance T Score
Description: Measurement: Self-reported measure of sleep disturbance, 90 days after surgery minus pre-intervention baseline Range: Standardized score with a mean of 50 and a standard deviation of 10 Interpretation: Higher scores indicate greater sleep disturbance
Time Frame: Between pre-intervention baseline and 90 days after surgery
Population: This was calculated in 22 patients who initiated the intervention and had the 90-day measurement after surgery.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 22
score on a scale | -3.0 [-4.7 to -1.3]

13. Other Pre Specified Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS)-Computer Adaptive Test (CAT) Social Roles/Activities Participation T Score
Description: Measurement: Self-reported measure of participation in social roles/activities, 90 days after surgery minus pre-intervention baseline Range: Standardized score with a mean of 50 and a standard deviation of 10 Interpretation: Higher scores indicate greater participation in social roles/activities
Time Frame: Between pre-intervention baseline and 90 days after surgery
Population: This was calculated in 22 patients who initiated the intervention and had the 90-day measurement after surgery.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 22
score on a scale | 1.6 [0.2 to 3.5]

14. Other Pre Specified Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS)-Computer Adaptive Test (CAT) Pain Interference T Score
Description: Measurement: Self-reported measure of pain interference, 90 days after surgery minus pre-intervention baseline Range: Standardized score with a mean of 50 and a standard deviation of 10 Interpretation: Higher scores indicate greater pain interference
Time Frame: Between pre-intervention baseline and 90 days after surgery
Population: This was calculated in 22 patients who initiated the intervention and had the 90-day measurement after surgery.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 22
score on a scale | -6.1 [-7.7 to -4.5]

15. Other Pre Specified Outcome: Change in Patient Reported Outcome Measurement Information System (PROMIS)-Computer Adaptive Test (CAT) Pain Intensity Score
Description: Measurement: Self-reported measure of pain intensity, 90 days after surgery minus pre-intervention baseline Range: 0 to 10 Interpretation: Higher scores indicate greater pain intensity
Time Frame: Between pre-intervention baseline and 90 days after surgery
Population: This was calculated in 22 patients who initiated the intervention and had the 90-day measurement after surgery.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 22
score on a scale | -1.4 [-1.8 to -1.1]

16. Other Pre Specified Outcome: 3-D Confusion Assessment Method
Description: Measurement: percentage of patients who develop delirium according to 3-D Confusion Assessment Method within 3 days of surgery
Time Frame: Between postoperative day 1 and day 3
Population: This was calculated in 23 patients who initiated the intervention and underwent surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prehabilitation
Number analyzed (Participants) | 23
Participants | 0

17. Other Pre Specified Outcome: Comprehensive Complication Index
Description: Measurement: a composite complication grading system by Clavien-Dindo Classification (CDC) after an intervention Range: 0 (no complications) to 100 (death) Interpretation: Higher scores indicate more severe complications
Time Frame: 1 month after surgery
Population: This was calculated in 23 patients who initiated the intervention and underwent surgery.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Prehabilitation
Number analyzed (Participants) | 23
score on a scale | 8.7 [0 to 25.7]

18. Other Pre Specified Outcome: Length of Stay
Description: Measurement: Number of hospital days from surgery until discharge
Time Frame: Between surgery and 1 month after surgery
Population: This was calculated in 23 patients who initiated the intervention and underwent surgery.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Prehabilitation
Number analyzed (Participants) | 23
days | 2 [2 to 3]

19. Other Pre Specified Outcome: 30-day Readmission From All Causes
Description: Measurement: percentage of patients who were readmitted within 30 days of surgery
Time Frame: Between surgery and 1 month after surgery
Population: This was calculated in 23 patients who initiated the intervention and underwent surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prehabilitation
Number analyzed (Participants) | 23
Participants | 3

20. Other Pre Specified Outcome: 30-day Mortality From All Causes
Description: Measurement: proportion of patients who died within 30 days of surgery
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Prehabilitation
Number analyzed (Participants) | 23
Participants | 0

21. Other Pre Specified Outcome: 90-day Mortality From All Causes
Description: Measurement: percentage of patients who died within 90 days of surgery
Time Frame: Between surgery and 90 days after surgery
Population: This was calculated in 23 patients who initiated the intervention and underwent surgery.
Measure: Count of Participants; unit: Participants
Arm/Group | Prehabilitation
Number analyzed (Participants) | 23
Participants | 1

22. Secondary Outcome: Adverse Events
Description: Measurement: percentage of patients who experience any adverse events per self-report Range: 0-100% (higher values indicate more adverse events)
Time Frame: Between pre-intervention baseline and post-intervention (up to 4 weeks)
Population: This was calculated in 28 patients who initiated the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Prehabilitation
Number analyzed (Participants) | 28
Participants | 8

ADVERSE EVENTS:
Time Frame: From enrollment until 90 days post-surgery
Description: Note: Adverse events and all-cause mortality were collected from 28 participants who initiated the intervention. Postoperative outcomes were collected from 23 participants who underwent surgery.
Arm/Group | Prehabilitation
All-Cause Mortality (participants affected / at risk) | 1/28
Serious Adverse Events (participants affected / at risk) | 1/28
Other Adverse Events (participants affected / at risk) | 7/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prehabilitation (N=28)
Esophageal bleeding (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prehabilitation (N=28)
Gastrointestinal discomforts (Gastrointestinal disorders) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The absence of a control group without prehabilitation does not allow evaluation of the intervention effect. The prehabilitation program was delivered by a clinical team with extensive experience in geriatric care. The feasibility in our study may not generalize to patients treated at other hospitals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT05752474/Prot_SAP_001.pdf